CLINICAL TRIAL: NCT00239889
Title: Efficacy and Safety of Salmon Calcitonin Nasal Spray in Improving Muscle Strength and Reducing Pain After Forearm Fracture in Postmenopausal Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CSMC051A2402
Record Dates: First submitted 2005-10-13; First posted 2005-10-17 (Estimated); Last update posted 2006-11-30 (Estimated); Status verified 2006-03

CONDITIONS: Forearm Fracture
Keywords: Forearm fracture; Postmenopausal women; Pain; Grip strength; Salmon calcitonin
MeSH Terms: conditions — Pain | interventions — salmon calcitonin

INTERVENTIONS:
Drug: Salmon calcitonin

SUMMARY:
Calcitonin has been used for many years for treating osteoporosis in postmenopausal women, and it has been shown that calcitonin reduces pain after spine and hip fracture in women with osteoporosis. Therefore, this study assesses the safety and efficacy of salmon calcitonin nasal spray on muscle strength after a forearm fracture, pain, quality of life and fracture healing in postmenopausal women.

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal women, aged at least 60 years old
* Having a forearm fracture within the last 3-7 days before treatment
* Fracture is treated with either a plaster cast only, or a cast plus Kirschner wires

Exclusion Criteria:

* Multiple fractures, severe fractures, or the forearm fractured in more than one place
* Nerve damage in the forearm caused by the fracture
* Other conditions which would interfere with the grip strength measurements (e.g. swelling, paralysis, skin diseases or rheumatoid arthritis)

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2002-03

PRIMARY OUTCOMES:
Grip strength of the injured arm after 24 weeks

SECONDARY OUTCOMES:
Post fracture pain intensity at rest in the evenings and analgesic consumption over 24 hours at Days 1-7; weeks 2, 3 and 4; the day before cast removal; 1 to 7 days and 2, 4 and 10 weeks after cast removal; and at 24 weeks after enrolment.
Post fracture pain intensity after grip strength assessment at cast removal; at 1, 2, 4 and 10 weeks after cast removal (4-6 weeks after fracture); and at 24 weeks after enrolment.
Incidence of complex regional pain syndrome (CRPS) type 1/reflex sympathetic dystrophy (RSD) at cast removal; at 1, 2, 4 and 10 weeks after cast removal; and at 24 weeks after enrolment.
Grip strength in the injured arm at cast removal and at 1, 2, 4 and 10 weeks after cast removal.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Basel 41 61 324 1111, Study Chair — Novartis
Locations (2):
- Novartis, Nuremberg, Germany
- Novartis, Basel, Switzerland